CLINICAL TRIAL: NCT05666102
Title: Transgender Men's Perspectives on HIV Risk and HIV Prevention
Brief Title: Transgender Men's Perspectives on HIV Risk and HIV Prevention Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Ricky Hill, Research Assistant Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STU00217158
Record Dates: First submitted 2022-11-21; First posted 2022-12-27 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Transgenderism; HIV Infections
Keywords: Transgender; LGBTQ; HIV; Qualitative
MeSH Terms: conditions — Transsexualism; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Focus Groups (Other): Focus groups will occur during the course of the study period.
  Interventions: Behavioral: Transgender men's perspectives on HIV risk and HIV prevention interventions

INTERVENTIONS:
Behavioral: Transgender men's perspectives on HIV risk and HIV prevention interventions — Investigators will enroll 30 TMSM in 5 focus groups where they will examine the unique contexts in which risk for HIV acquisition occurs for TMSM, and explore participant preferences for HIV prevention services. Focus group questions will focus on five areas: 1) Gathering information related to partner selection and sorting among TMSM; 2) assessing TMSM's perceptions of HIV risk in their lived experiences; 3) exploring the various types of sexual behavior TMSM are engaging in; 4) understanding the various HIV prevention strategies currently being deployed by TMSM; and 5) examine the preferences TMSM have for receiving information related to sexual health and HIV prevention information.

SUMMARY:
The goal of this pilot study is to gather and analyze qualitative data from focus groups with Transgender men who have sex with men (TMSM) to learn more about the life experiences unique to TMSM that influence their attitudes and beliefs about HIV risk, as well as to better understand the intersections of these specific sexual and gender identities.

DETAILED DESCRIPTION:
Men who have sex with men (MSM) are disproportionately impacted by HIV in the United States. While most new HIV infections are assumed to occur between cisgender men who have sex with other cisgender men, an increasing body of literature proposes that transgender men and transmasculine people who have sex with cisgender men (TMSM) might be at elevated risk for HIV infection. Despite data suggesting that transgender men and cisgender men are regularly engaging in sexual relationships, the majority of research on HIV among MSM focuses almost exclusively on sexual partnerships between cisgender gay and bisexual men. Additionally, when HIV prevention research does include transgender people, it almost exclusively focuses on HIV risk within transgender women and transfeminine people. TMSM are rarely mentioned as potential sexual partners for cisgender men and have historically been left out of most research on HIV prevention and in preventive intervention development. The goal of this pilot study is to gather and analyze qualitative data from focus groups with TMSM to learn more about the life experiences unique to TMSM influence their attitudes and beliefs about HIV risk, as well as to better understand the intersections of these specific sexual and gender identities. The investigators will enroll 30 TMSM in 5 focus groups where they will examine the unique contexts in which risk for HIV acquisition occurs for TMSM, and explore participant preferences for HIV prevention services. Focus group questions will focus on five areas: 1) Gathering information related to partner selection and sorting among TMSM; 2) assessing TMSM's perceptions of HIV risk in their lived experiences; 3) exploring the various types of sexual behavior TMSM are engaging in; 4) understanding the various HIV prevention strategies currently being deployed by TMSM; and 5) examine the preferences TMSM have for receiving information related to sexual health and HIV prevention information. Focus group guide content areas may be updated in subsequent groups to reflect additional topics that may emerge from conversations in prior focus groups. Data from the groups will be analyzed by the investigator and study team using an iterative, thematic process. These themes will be synthesized in the development of culturally relevant HIV prevention interventions for TMSM.

ELIGIBILITY:
Inclusion Criteria:

* 18+; living in the United States;
* Assigned female at birth;
* Current gender identity of trans man or transmasculine;
* Sexual orientation of NOT heterosexual;
* Has access to the Internet.

Exclusion Criteria:

* Under 18;
* Living outside of the US;
* Assigned male at birth;
* Current gender identity OUTSIDE of transgender man or transmasculine person;
* Heterosexual/straight;
* Does not have access to the Internet.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Study is open to individuals assigned/designated female at birth (AFAB/DFAB) but who currently identify as a transgender man or transmasculine person.
Enrollment: 38 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Post-hoc thematic analysis across five domains | up to 9 months
  Post-focus group thematic analysis of attitudes and preferences of HIV prevention messaging and strategies for transgender men and transmasculine people in five separate domains:
  1. Partner selection and sorting among trans men who have sex with cis men (TMSM);
  2. TMSM's perceptions of HIV risk in their lived experiences;
  3. Exploring the various types of sexual behavior TMSM are engaging in;
  4. Understanding HIV prevention strategies currently used by TMSM; and
  5. Examine the preferences TMSM have for receiving information related to sexual health and HIV prevention.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Sexual and Gender Minority Health and Wellbeing, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT05666102/ICF_000.pdf